CLINICAL TRIAL: NCT02477475
Title: NEXIUM Capsule Specific Clinical Experience Investigation (S-CEI) to Investigate Treatment Response to NEXIUM in Patients With Reflux Esophagitis (RE) - Justification of Esomeprazole in Acid Related Disease for Reflux Symptom Healing Based on Patient Clinical Outcomes
Brief Title: Nexium Capsules S-CEI for Justification of Esomeprazole in Acid Related Disease for Reflux Symptom Healing Based on Patient Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961HL00020
Record Dates: First submitted 2015-06-18; First posted 2015-06-22 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Reflux Esophagitis
Keywords: reflux esophagitis; Nexium
MeSH Terms: conditions — Esophagitis, Peptic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NEXIUM: Oral dose 20mg/day

SUMMARY:
The objective of this investigation is to collect following data in patients given NEXIUM capsule (NEXIUM) in usual post-marketing use.

DETAILED DESCRIPTION:
Primary objective To investigate treatment response to NEXIUM in patients with reflux esophagitis (RE).

Secondary objectives

To investigate following items in patients with RE:

1. Patient satisfactory level of the treatment for RE
2. Health-related quality of life (HRQOL)
3. Severity and frequency of RE symptoms reported by physicians
4. Endoscopic healing rate
5. Development of ADRs

ELIGIBILITY:
Inclusion Criteria:

* Patients to be enrolled in this S-CEI must fulfill all the criteria below at the start of the treatment with NEXIUM.

  1. Aged at least 20 years.
  2. Patients who has a current or past history of clinically diagnosed RE
  3. Patients whose answers in the baseline GerdQ include "2-3 days" or "4-7 days" in at least one of the questions Nos 1, 2, 5 and 6.
  4. Patients to whom NEXIUM 20 mg once daily is to be administered for RE
  5. Patients from whom written consent has been obtained.

Exclusion Criteria:

* Patients must not enter the investigation if any of the following exclusion criteria are fulfilled at the start of the treatment with NEXIUM:

  1. Patients whose ability to follow instructions are suspected to be low by physicians
  2. Patients with a past history of hypersensitivity to the ingredients of NEXIUM.
  3. Patients receiving atazanavir sulfate or rilpivirine hydrochloride
  4. Patients who have received NEXIUM within the past eight weeks for treatment of RE

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Since the target patient population of the S-CEI is symptomatic RE patients, the patients fulfilling the inclusion criteria and not the exclusion criteria shown below will be enrolled as the subjects of this investigation.
Sampling Method: Non-Probability Sample
Enrollment: 1595 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
Treatment response to NEXIUM based on answers in GerdQ | at the time of Treatment Week 8
  The rate of patients whose answers in the GerdQ are "none" or "one day" in the questions Nos 1, 2, 5 and 6 at the end of the observation.
  GerdQ is a questionnaire for assessment of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — AstraZeneca
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: AZ_Synopsis_D961HL00020_STUDY_REPORT_SUMMARY — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3915&filename=AZ_Synopsis_D961HL00020_STUDY_REPORT_SUMMARY.pdf